CLINICAL TRIAL: NCT04228770
Title: Pharmacist-led Perioperative Medicines Optimisation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PH18/112828
Record Dates: First submitted 2020-01-10; First posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Pharmacists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Warfarin patients (Experimental): Patients on high risk medication - warfarin
  Interventions: Behavioral: Meeting with pharmacist
- Parkinson's patients (Experimental): Patients with high risk disease - parkinson's
  Interventions: Behavioral: Meeting with pharmacist

INTERVENTIONS:
Behavioral: Meeting with pharmacist — Meeting with pharmacist to support drug management following their routine surgery.

SUMMARY:
Patients attend pre-assessment clinics (POAC) who require an elective operation and who are having a general anaesthetic. At POAC patients are asked about their health, and past medical conditions to assess their fitness for anaesthetic, a list of medicines taken is documented. Patients can then be given a date for surgery. During their stay in hospital patients will see a pharmacist who confirms what medicines are being taken, and ensures those medicines are prescribed and available during the patients stay.

This study is aimed at improving the care of patients who are admitted for elective surgery. The study will review two different interventions made prior to a patient's admission for surgery. One will look at a group of patients taking a high risk medicine and the other a group of patients with a high risk disease. The high risk medicine chosen is warfarin, and the high risk disease is Parkinson's disease. It is known that inappropriate or lack of medicines management in these groups can result in delayed surgery, poorer surgical outcomes and can affect a patient's recovery after surgery. Due to patient numbers and the variability between patients being too great, and a lack of research in this area a controlled trial cannot be performed. This complex intervention will review the interventions made, to understand how and why the interventions change care and what it is specifically within the interventions that are exerting a positive effect to improve care. All elective surgical patients who attend POAC at St James' University Hospital who are either, taking warfarin or who have Parkinson's disease will be seen by a pharmacist. An accurate drug history will be taken and if changes are required to medications these will be resolved at the POAC appointment. Patients will be provided with an individualised perioperative medication plan.

ELIGIBILITY:
Inclusion Criteria:

* Participant has capacity.
* Participants must be attending the POAC at St James' University Hospital
* Scheduled elective surgery or other procedures requiring general anaesthesia
* Male or Female, aged 18 years or above.
* Diagnosed with Parkinson's Disease or taking warfarin
* In the Investigator's opinion, is able and willing to comply with all requirements of the intervention.

Exclusion Criteria:

* Female participant who is pregnant, lactating or planning pregnancy during the course of the intervention.
* Under 17years of age
* Participants who are having a local anaesthetic
* Any who are having emergency surgery
* Participants who are unable to provide consent
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk or may influence the result, or the participant's ability to participate in the intervention.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-01-10 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Interview with Pharmacist | 1 hour
  Interview with Pharmacist to support the management of the patients drug regime

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospital NHS Trust, Leeds, United Kingdom